CLINICAL TRIAL: NCT01483989
Title: In Vivo Measurement of Corneal Epithelial Changes in Dry Eye(DE) Patients
Brief Title: In Vivo Measurement of Corneal Epithelial Changes in Dry Eye Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-49
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye; Epithelial changes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYSTANE® Gel Drops Lubricant eye gel (Experimental): SYSTANE Gel Drops Lubricant Eye gel dosed (bilaterally) 3 times per day for the 28 day period.
  Interventions: Other: SYSTANE® Gel Drop lubricant eye gel

INTERVENTIONS:
Other: SYSTANE® Gel Drop lubricant eye gel — SYSTANE Gel Drops Lubricant Eye gel dosed (bilaterally) 3 times per day for the 28 day period.
  Other Names: Systane Gel

SUMMARY:
The purpose of this study is to measure corneal epithelial changes in dry eye subjects using a novel lubricant eye gel.

DETAILED DESCRIPTION:
The purpose of this study is to measure corneal epithelial changes in dry eye (DE) subjects using a novel lubricant eye gel.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have history of dry eye as determined by:

1. Questionnaire
2. Tear Film Break Up Time less than or equal to 10 seconds
3. Schirmer's score of less than or equal to 5 mm
4. Corneal staining greater than or equal to 3 in either eye, and
5. Positive for conjunctival staining (greater than or equal to 1)

Exclusion Criteria:

* Patients cannot wear contact lenses within 1 week prior nor during the study, and cannot have a history of hypersensitivity to any component of Systane Gel Drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes in epithelial irregularity following 4 weeks of treatment with a novel artificial tear gel. | baseline and 28 days
  The Changes in epithelial irregularity following 4 weeks of treatment with a novel artificial tear gel.

REFERENCES:
- [Result] http://iovs.arvojournals.org/article.aspx?articleid=2351788